CLINICAL TRIAL: NCT06101979
Title: A Prospective Study of Fortiva in Hernia Repair
Status: Enrolling by invitation | Type: Observational
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: RTI-2022-01
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Ventral Hernia; Incisional Hernia; Abdominal Wall Reconstruction
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fortiva Tissue Matrix
  Interventions: Device: Fortiva Tissue Matrix

INTERVENTIONS:
Device: Fortiva Tissue Matrix — Acellular Dermal Matrix used in hernia surgery

SUMMARY:
The goal of this study is to evaluate safety and performance of the Fortiva Tissue Matrix. Participants will complete questionnaires to measure outcomes after hernia surgery for two years.

DETAILED DESCRIPTION:
This is a post market, prospective, multi-center study of up to 120 participants at approximately 10 clinical study sites. Safety and performance will be measured after hernia repair for two years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age at time of consent
* Undergoing hernia surgery in which Fortiva Tissue Matrix will be used
* Have no contraindications to the test material (s)
* Able to provide informed consent
* Able to read, understand and complete study questionnaires
* Able and willing to return for scheduled study visits

Exclusion Criteria:

* <18 years of age
* American Society of Anesthesiologists (ASA) physical class of 4,5 or 6
* Currently enrolled or plans to enroll in another clinical study that would affect the validity of the study
* Hernia repairs involving active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be candidates for hernia surgery recruited from the participating Investigator's population
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Type of adverse events | 6 weeks, 6 months, 12 months and 24 months

SECONDARY OUTCOMES:
Patient satisfaction | 6 weeks, 6 months, 12 months and 24 months
  SF-36 questionnaire has 8 multi-item scales with a higher score representing better health status. Each domain has a score range of 0-100
Pain measured using the visual analog scale for pain | 6 weeks, 6 months, 12 months and 24 months
  Visual Analog Scale using a scale of 0-10 with 0 being no pain and 10 being unbearable pain
Implant failure | 6 weeks, 6 months, 12 months and 24 months
  Partial or total removal of Fortiva Tissue Matrix
Hernia recurrence | 12 months
  Hernia recurrence requiring surgical reintervention

CONTACTS AND LOCATIONS:
Locations (1):
- James Paget University Hospital, Great Yarmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No